CLINICAL TRIAL: NCT01668212
Title: Perifollicular Doppler in Natural Cycle In Vitro Fertilization
Status: Completed | Type: Observational
Sponsor: Clinique Ovo (Industry)
Responsible Party: Sponsor
Other Study IDs: OVO-11-01
Record Dates: First submitted 2012-06-19; First posted 2012-08-20 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- natural In Vitro Fertilization cycle: Patient doing following natural In Vitro fertilization cycle
  Interventions: Procedure: Doppler ultrasound

INTERVENTIONS:
Procedure: Doppler ultrasound — Doppler Ultrasound

SUMMARY:
Perifollicular Doppler could reflect the quality of the follicle's vascularization and, consequently, the one of the oocyte that ensues from it. Perifollicuar Doppler is the analysis, in ultrasound, of the blood flow in vessels surrounding the follicle.

The goal of this study is to evaluate if there is a link, in natural cycle In Vitro Fertilization, between the quality of the vascularization and the one of the oocyte, the embryo and the pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a natural In Vitro Fertilization cycle.
* Patient under 38 years old
* Body mass indice under 35
* Ovulatory cycles between 20-35 days

Exclusion Criteria:

* Patient with a stimulation In Vitro Fertilization cycle
* Patient with a naturalIn Vitro Fertilization cycle with egg donor
* Patient with a natural In Vitro Fertilization cycle with freezing embryo
* Smoking patient
* Diabetic patient
* Patient with treatment of antihypertensive drug, anticoagulant, antiplatelet, vasodilator
* Body mass indice over 35
* Patient over 38 years old
* Patient without ovulation or cycle over 35 days
* Percutaneous Epididymal Sperm Aspiration (PESA), Testicular Sperm Extraction (TESE) or micro TESE

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women following In Vitro Fertilization cycle
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2012-03; Primary Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Quality perifollicular doppler and quality of the oocyte | 2 weeks
  The measurements are done twice; on days of induction and oocyte retrieval. During the blood sample collection on the day of the induction, there is also a measurement of progesterone, estradiol and luteinizing hormone (LH).

CONTACTS AND LOCATIONS:
Overall Officials: Delphine Delrieu, MD, Principal Investigator — Clinique Ovo
Locations (1):
- Ovo Fertilité, Montreal, Quebec, Canada